CLINICAL TRIAL: NCT05764902
Title: Interventions to Reduce Loneliness in Elderly Patients in the Cardiac ICU (CICU): A Randomized Control Trial
Brief Title: Interventions to Reduce Loneliness in Elderly Patients in the Cardiac ICU (CICU)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poriya Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0079-19-POR
Record Dates: First submitted 2023-02-17; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Loneliness
Keywords: Intensive Care Units; Older Adult; Aged

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial will evaluate the impact of tailored interventions on loneliness levels of patients admitted to the Cardiac ICU (CICU) at the Baruch Padeh Poriya Medical Center. A questionnaire using a 12-point Likert scale, adapted from the University of California Los Angeles (UCLA) and De Jong Gierveld Loneliness Scales, will be used to assess loneliness levels at CICU admission and discharge. Patients will be randomized into the intervention or control group. The intervention group will receive an additional questionnaire to assess their individual needs and preferences. CICU staff will provide individualized interventions to address the expressed needs and preferences of the intervention group, while the control group will receive standard care. Changes in loneliness levels during CICU hospitalization will be compared between the groups.
Who Masked: Outcomes Assessor
Masking Description: The assessors who analyze the data will be blinded to the allocation of patients to the intervention or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients will receive standard of care.
- Intervention (Experimental): The intervention group will be given an additional questionnaire assessing individual needs and preferences. CICU staff will provide patient-tailored interventions based on the expressed needs and preferences of those in the intervention group.
  Interventions: Behavioral: Patient-tailored intervention

INTERVENTIONS:
Behavioral: Patient-tailored intervention — The intervention group will receive various tailored interventions designed to address multiple patient preferences, including sleeping, eating, and resting habits, hobbies, visitation preferences, religious and spiritual needs, preferences for independence and privacy, and any other specific requests or requirements.
  Arms: Intervention

SUMMARY:
This clinical trial aims to study whether patient-tailored interventions can reduce loneliness levels in elderly patients admitted to the Cardiac ICU (CICU). The study will involve an experimental group that will receive tailored interventions based on their needs and preferences, and a control group that will receive standard care. The primary goal of the trial is to determine if patient-tailored interventions can effectively reduce loneliness in patients staying in the CICU. The trial is interventional in nature and will compare results between the two groups.

DETAILED DESCRIPTION:
This interventional clinical trial is designed to investigate the effects of patient-tailored interventions on reducing loneliness levels in elderly patients admitted to the Cardiac ICU (CICU). The aim of this study is to determine if tailored interventions can improve the well-being and quality of life of elderly patients who experience loneliness during their stay in the hospital.

The primary research question is: Could patient-tailored interventions be used to reduce loneliness in patients staying in the CICU? The study will involve two groups of participants: an experimental group that will receive tailored interventions and a control group that will receive standard care.

Participants in the experimental group will receive tailored interventions by CICU staff based on their expressed needs and preferences. The interventions will be personalized to the individual patient and will be individualized based on survey responses from patients in the experimental group. The interventions will be implemented throughout the patient's stay in the CICU.

The control group will receive standard care, which includes medical treatment and monitoring, but will not receive any patient-tailored interventions aimed at reducing loneliness levels.

ELIGIBILITY:
Inclusion Criteria:

* patients who were able to communicate effectively and cooperate with staff members
* patients who had stayed in the CICU for a minimum of 48 hours
* patients who met the age criteria of being over 70 years old

Exclusion Criteria:

* patients under the age of 70 years old
* patients who were unconscious or on ventilators
* patients who were admitted immediately after surgery
* patients with hemodynamic and/or respiratory instability
* patients with cognitive impairments, such as dementia and/or Alzheimer's disease

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-28 (Actual); Primary Completion 2023-03-10 (Estimated); Study Completion 2023-05-10 (Estimated)

PRIMARY OUTCOMES:
Loneliness levels | Reduction in loneliness levels will be assessed at baseline and weekly during the patient's stay in the CICU until immediately before discharge, for a total of 4 weeks.
  We developed a 12-item self-reported questionnaire by adapting questions from two established loneliness scales: the De Jong Gierveld Loneliness Scale and the UCLA Loneliness Scale. Two unique questions were also included in the survey. Each item was rated on a 5-point Likert scale. Total loneliness scores ranged from 12 to 60, with higher scores indicating greater loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Erez Kachel, MD, Study Director — Poriya Medical Center
Locations (1):
- Baruch Padeh (Poriya) Medical Center, Poria – Neve Oved, Israel

REFERENCES:
- [Background] Perissinotto CM, Stijacic Cenzer I, Covinsky KE. Loneliness in older persons: a predictor of functional decline and death. Arch Intern Med. 2012 Jul 23;172(14):1078-83. doi: 10.1001/archinternmed.2012.1993. PMID 22710744
- [Background] Holt-Lunstad J, Smith TB, Baker M, Harris T, Stephenson D. Loneliness and social isolation as risk factors for mortality: a meta-analytic review. Perspect Psychol Sci. 2015 Mar;10(2):227-37. doi: 10.1177/1745691614568352. PMID 25910392
- [Background] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660
- [Background] Adepoju OE, Chae M, Woodard L, Smith KL, Herrera L, Han D, Howard DL, Dobbins J, Ory M. Correlates of Social Isolation Among Community-Dwelling Older Adults During the COVID-19 Pandemic. Front Public Health. 2021 Dec 10;9:702965. doi: 10.3389/fpubh.2021.702965. eCollection 2021. PMID 34956998
- [Background] Ernst M, Niederer D, Werner AM, Czaja SJ, Mikton C, Ong AD, Rosen T, Brahler E, Beutel ME. Loneliness before and during the COVID-19 pandemic: A systematic review with meta-analysis. Am Psychol. 2022 Jul-Aug;77(5):660-677. doi: 10.1037/amp0001005. Epub 2022 May 9. PMID 35533109
- [Background] National Academies of Sciences, Engineering, and Medicine; Division of Behavioral and Social Sciences and Education; Health and Medicine Division; Board on Behavioral, Cognitive, and Sensory Sciences; Board on Health Sciences Policy; Committee on the Health and Medical Dimensions of Social Isolation and Loneliness in Older Adults. Social Isolation and Loneliness in Older Adults: Opportunities for the Health Care System. Washington (DC): National Academies Press (US); 2020 Feb 27. Available from http://www.ncbi.nlm.nih.gov/books/NBK557974/ PMID 32510896
- [Background] Hawkley LC, Cacioppo JT. Loneliness matters: a theoretical and empirical review of consequences and mechanisms. Ann Behav Med. 2010 Oct;40(2):218-27. doi: 10.1007/s12160-010-9210-8. PMID 20652462
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Cacioppo JT, Hawkley LC, Thisted RA. Perceived social isolation makes me sad: 5-year cross-lagged analyses of loneliness and depressive symptomatology in the Chicago Health, Aging, and Social Relations Study. Psychol Aging. 2010 Jun;25(2):453-63. doi: 10.1037/a0017216. PMID 20545429
- [Background] Hawkley LC, Preacher KJ, Cacioppo JT. Loneliness impairs daytime functioning but not sleep duration. Health Psychol. 2010 Mar;29(2):124-9. doi: 10.1037/a0018646. PMID 20230084
- [Background] Hawkley LC, Thisted RA, Cacioppo JT. Loneliness predicts reduced physical activity: cross-sectional & longitudinal analyses. Health Psychol. 2009 May;28(3):354-63. doi: 10.1037/a0014400. PMID 19450042
- [Background] Wilson RS, Krueger KR, Arnold SE, Schneider JA, Kelly JF, Barnes LL, Tang Y, Bennett DA. Loneliness and risk of Alzheimer disease. Arch Gen Psychiatry. 2007 Feb;64(2):234-40. doi: 10.1001/archpsyc.64.2.234. PMID 17283291
- [Background] Cacioppo S, Grippo AJ, London S, Goossens L, Cacioppo JT. Loneliness: clinical import and interventions. Perspect Psychol Sci. 2015 Mar;10(2):238-49. doi: 10.1177/1745691615570616. PMID 25866548
- [Background] Masi CM, Chen HY, Hawkley LC, Cacioppo JT. A meta-analysis of interventions to reduce loneliness. Pers Soc Psychol Rev. 2011 Aug;15(3):219-66. doi: 10.1177/1088868310377394. Epub 2010 Aug 17. PMID 20716644
- [Background] Fakoya OA, McCorry NK, Donnelly M. Loneliness and social isolation interventions for older adults: a scoping review of reviews. BMC Public Health. 2020 Feb 14;20(1):129. doi: 10.1186/s12889-020-8251-6. PMID 32054474
- [Background] Boekhout JM, Volders E, Bolman CAW, de Groot RHM, Lechner L. Long-Term Effects on Loneliness of a Computer-Tailored Intervention for Older Adults With Chronic Diseases: A Randomized Controlled Trial. J Aging Health. 2021 Dec;33(10):865-876. doi: 10.1177/08982643211015027. Epub 2021 May 7. PMID 33962517
- [Background] Luo Y, Hawkley LC, Waite LJ, Cacioppo JT. Loneliness, health, and mortality in old age: a national longitudinal study. Soc Sci Med. 2012 Mar;74(6):907-14. doi: 10.1016/j.socscimed.2011.11.028. Epub 2012 Jan 25. PMID 22326307
- [Background] Valtorta N, Hanratty B. Loneliness, isolation and the health of older adults: do we need a new research agenda? J R Soc Med. 2012 Dec;105(12):518-22. doi: 10.1258/jrsm.2012.120128. No abstract available. PMID 23288086
- [Background] Czaja SJ, Boot WR, Charness N, Rogers WA, Sharit J. Improving Social Support for Older Adults Through Technology: Findings From the PRISM Randomized Controlled Trial. Gerontologist. 2018 May 8;58(3):467-477. doi: 10.1093/geront/gnw249. PMID 28201730
- [Background] Gardiner C, Geldenhuys G, Gott M. Interventions to reduce social isolation and loneliness among older people: an integrative review. Health Soc Care Community. 2018 Mar;26(2):147-157. doi: 10.1111/hsc.12367. Epub 2016 Jul 13. PMID 27413007
- [Background] Knox SS, Uvnas-Moberg K. Social isolation and cardiovascular disease: an atherosclerotic pathway? Psychoneuroendocrinology. 1998 Nov;23(8):877-90. doi: 10.1016/s0306-4530(98)00061-4. PMID 9924742
- [Background] Williams CYK, Townson AT, Kapur M, Ferreira AF, Nunn R, Galante J, Phillips V, Gentry S, Usher-Smith JA. Interventions to reduce social isolation and loneliness during COVID-19 physical distancing measures: A rapid systematic review. PLoS One. 2021 Feb 17;16(2):e0247139. doi: 10.1371/journal.pone.0247139. eCollection 2021. PMID 33596273
- [Background] Russell DW. UCLA Loneliness Scale (Version 3): reliability, validity, and factor structure. J Pers Assess. 1996 Feb;66(1):20-40. doi: 10.1207/s15327752jpa6601_2. PMID 8576833
- [Background] De Jong Gierveld J, Van Tilburg T. The De Jong Gierveld short scales for emotional and social loneliness: tested on data from 7 countries in the UN generations and gender surveys. Eur J Ageing. 2010 Jun;7(2):121-130. doi: 10.1007/s10433-010-0144-6. Epub 2010 Apr 9. PMID 20730083